CLINICAL TRIAL: NCT01945294
Title: A Phase 3 Clinical Trial to Study Short Duration Versus Standard Response-Guided Therapy With MK-3034 (SCH 503034)/Boceprevir Combined With PegIntron and Ribavirin in Previously Untreated Non-Cirrhotic Subjects With Chronic HCV Genotype 1 in Asia
Brief Title: Short Duration Versus Standard Response-Guided Therapy With Boceprevir Combined With PegIntron and Ribavirin in Previously Untreated Non-Cirrhotic Asian Participants With Chronic HCV Genotype 1 (MK-3034-107)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3034-107
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: 16-week Treatment Arm (Experimental): All screened and enrolled participants initially underwent a 12-week (4 weeks PR + 8 weeks BOC + PR) lead-in treatment period prior to randomization to Arms 1 or 2 (participants with undetectable HCV RNA) or allocation to Arm 3 (participants with detectable HCV RNA). After completing the 12-week lead-in, participants with undetectable HCV RNA were randomized to receive an additional 4 weeks of BOC + PR, for a total of 16 weeks of treatment. At Week 16, participants underwent 12 weeks of follow-up (participation complete at Week 28).
  Interventions: Drug: Boceprevir; Biological: Peg-interferon alfa-2b; Drug: Ribavirin
- Arm 2: 28-week Treatment Arm (Experimental): All screened and enrolled participants initially underwent a 12-week (4 weeks PR + 8 weeks BOC + PR) lead-in treatment period prior to randomization to Arms 1 or 2 (participants with undetectable HCV RNA) or allocation to Arm 3 (participants with detectable HCV RNA). After completing the 12-week lead-in, participants with undetectable HCV RNA were randomized to receive an additional 16 weeks of BOC + PR, for a total of 28 weeks of treatment. At Week 28, participants underwent 12 weeks of follow-up (participation complete at Week 40).
  Interventions: Drug: Boceprevir; Biological: Peg-interferon alfa-2b; Drug: Ribavirin
- Arm 3: 48-week Treatment Arm (Experimental): All screened and enrolled participants initially underwent a 12-week (4 weeks PR + 8 weeks BOC + PR) lead-in treatment period prior to randomization to Arms 1 or 2 (participants with undetectable HCV RNA) or allocation to Arm 3 (participants with detectable HCV RNA). After completing the 12-week lead-in, participants with detectable HCV RNA were allocated to receive an additional 24 weeks of BOC + PR and an additional 12 weeks of PR, for a total of 48 weeks of treatment. At Week 48, participants underwent 12 weeks of follow-up (participation complete at Week 60).
  Interventions: Drug: Boceprevir; Biological: Peg-interferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Drug: Boceprevir — 800 mg three times daily orally
  Other Names: MK-3034
Biological: Peg-interferon alfa-2b — 1.5 mcg/kg weekly subcutaneously
  Other Names: PegIntron
Drug: Ribavirin — 800-1400 mg twice-daily divided orally based on body weight
  Other Names: Rebetol

SUMMARY:
The purpose of this study is to estimate the difference in the efficacy between a 16-week treatment regimen of boceprevir (BOC) in combination with peg-intron alpha 2b (P) plus ribavirin (R) (BOC + PR) and a 28-week treatment regimen of BOC + PR in previously untreated participants with chronic hepatitis C (CHC) genotype 1 in Asia who achieve undetectable hepatitis C virus ribonucleic acid (HCV RNA).

ELIGIBILITY:
Inclusion Criteria:

* weigh ≥ 40 kg and ≤ 125 kg
* have CHC genotype 1 infection
* has had a liver biopsy or non-invasive liver fibrosis test that shows no evidence of cirrhosis and hepatocellular carcinoma
* must agree that the participant and the participant's partner will each use acceptable methods of contraception for at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study medication, or longer if dictated by local regulations (for a female participant who is of childbearing potential or male participant with female sexual partner who is of childbearing potential)

Exclusion Criteria:

* participates in any other interventional clinical trial within 30 days of the screening visit in this trial or intends to participate in another interventional clinical trial during participation in this trial
* is co-infected with human immunodeficiency virus (HIV) or hepatitis B virus
* has evidence or history of chronic hepatitis not caused by HCV, including but not limited to nonalcoholic steatohepatitis (NASH), drug-induced hepatitis, and autoimmune hepatitis
* has evidence of decompensated liver disease including, but not limited to, a history or presence of clinical ascites, bleeding varices, or hepatic encephalopathy
* has evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC
* has evidence of active or suspected malignancy, or a history of malignancy, within the last 5 years
* has been previously treated with an interferon or ribavirin regimen or HCV direct acting anti-viral regimen, or treated for hepatitis C with any investigational medication
* taking/plans to take significant inducers of inhibitors of Cytochrome P450 3A4 (CYP3A4) substrates 2 weeks prior to start of study medications, or herbal supplements, including but not limited to St. John's Wort 2 weeks prior to start of study medications (Day 1)
* has pre-existing psychiatric condition(s)
* has a clinical diagnosis of substance abuse
* has any known medical condition that could interfere with the participation in and completion of the trial including immunologically-mediated disease, chronic pulmonary disease, or current or history of any clinically significant cardiac abnormalities/dysfunction
* is pregnant or nursing (for female participant) or female partner intends to become pregnant (for male participant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2015-08-05 (Actual); Study Completion 2015-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment-naïve adult male and female participants with chronic hepatitis C virus (HCV) genotype 1 (GT1) infection were recruited in the Asia-Pacific region.
Groups:
- All Treated Participants: All screened and enrolled participants initially underwent a 12-week (4 weeks PR + 8 weeks BOC + PR) lead-in treatment period prior to randomization to Arms 1 or 2 (participants with undetectable hepatitis C virus [HCV] ribonucleic acid [RNA]) or allocation to Arm 3 (participants with detectable HCV RNA).
- Arm 1: 16-week Treatment Arm: After completing the 12-week lead-in, participants with undetectable HCV RNA were randomized to receive an additional 4 weeks of BOC + PR, for a total of 16 weeks of treatment. At Week 16, participants underwent 12 weeks of follow-up (participation complete at Week 28).
- Arm 2: 28-week Treatment Arm: After completing the 12-week lead-in, participants with undetectable HCV RNA were randomized to receive an additional 16 weeks of BOC + PR, for a total of 28 weeks of treatment. At Week 28, participants underwent 12 weeks of follow-up (participation complete at Week 40).
- Arm 3: 48-week Treatment Arm: After completing the 12-week lead-in, participants with detectable HCV RNA were allocated to receive an additional 24 weeks of BOC + PR and an additional 12 weeks of PR, for a total of 48 weeks of treatment. At Week 48, participants underwent 12 weeks of follow-up (participation complete at Week 60).
Period: Period 1: 12-Week PR + BOC Lead-In
Arm/Group | All Treated Participants | Arm 1: 16-week Treatment Arm | Arm 2: 28-week Treatment Arm | Arm 3: 48-week Treatment Arm
Started | 257 | 0 | 0 | 0
Completed | 236 | 0 | 0 | 0
Not Completed | 21 | 0 | 0 | 0
Period: Period 2: BOC+ PR Treatment & Follow-up
Arm/Group | All Treated Participants | Arm 1: 16-week Treatment Arm | Arm 2: 28-week Treatment Arm | Arm 3: 48-week Treatment Arm
Started | 0 (Participants were assigned to 1 of the 3 arms after upon the 12-week BOC + PR lead-in.) | 102 | 105 | 29
Completed | 0 | 97 | 97 | 23
Not Completed | 0 | 5 | 8 | 6

BASELINE CHARACTERISTICS:
Population: The total number of participants in Arm 3 (i.e., n=50) includes participants who completed the BOC + PR lead-in and were allocated at Week 12 based on having detectable HCV RNA (n=29), as well as participants who began the BOC + PR lead-in but discontinued prior to Week 12 (n=21).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: 16-week Treatment Arm | Arm 2: 28-week Treatment Arm | Arm 3: 48-week Treatment Arm | Total
Number analyzed (Participants) | 102 | 105 | 50 | 257
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (11.1) | 44.6 (10.6) | 46.5 (11.8) | 44.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 41 | 24 | 108
  Male | 59 | 64 | 26 | 149

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Undetectable HCV RNA Who Achieve Sustained Viral Response at Follow-up Week 12 (SVR12) [16-Week Arm vs. 28-Week Arm]
Description: SVR12 was declared when participants who had undetectable HCV RNA (HCV RNA < Lower Limit of Quantification [LLoQ]) after the 12-week lead-in also had undetectable HCV RNA 12 weeks after completing their assigned BOC treatment regimen. The Roche COBAS™ Taqman™ automated HCV test (v2.0 assay) used in this study has a LLoQ of 15 IU/mL.
Time Frame: Follow-up Week (FW) 12 (up to 40 weeks)
Population: Participants of the Full Analysis Set (FAS) who were treated with any study medication, had undetectable HCV RNA at TW8, and were randomized to Arm 1 or Arm 2. Participants in Arm 3 were not included in the primary efficacy analysis as pre-specified by the protocol.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm 1: 16-week Treatment Arm | Arm 2: 28-week Treatment Arm | Arm 3: 48-week Treatment Arm
Number analyzed (Participants) | 102 | 105 | 0
Percentage of Participants | 70.6 | 81.9 |
Statistical Analysis 1: Comparison: Arm 1: 16-week Treatment Arm vs Arm 2: 28-week Treatment Arm; Test type: Superiority or Other; Difference in SVR12 percentage = -11.4, 95% CI 2-sided [-23.2 to 0.4]

2. Secondary Outcome: Percentage of Participants With Undetectable HCV RNA Across Treatment
Description: The percentage of participants with undetectable HCV RNA (HCV RNA <LLoQ) at TW4, TW8, and TW12 is summarized for each arm. The Roche COBAS™ Taqman™ automated HCV test (v2.0 assay) used in this study has a LLoQ of 15 IU/mL.
Time Frame: TW4, TW8, and TW12
Population: Participants in the FAS population (consisting of all participants treated with any study medication who had undetectable HCV RNA at TW8 and were randomized to Arm 1 or Arm 2, and participants with detectable HCV RNA at TW8 in Arm 3) with available data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm 1: 16-week Treatment Arm | Arm 2: 28-week Treatment Arm | Arm 3: 48-week Treatment Arm
Number analyzed (Participants) | 101 | 105 | 29
Percentage of Participants
  TW4 | 24.8 | 17.1 | 0.0
  TW8 | 100.0 | 100.0 | 0.0
  TW12 | 99.0 | 100.0 | 69.0

3. Secondary Outcome: Percentage of Participants Achieving SVR12 Among Participants With Undetectable HCV RNA Across Treatment
Description: The percentage of participants achieving SVR12 who had undetectable HCV RNA (HCV RNA <LLoQ) at Week 4, Week 8, and Week 12 is summarized for each arm. The Roche COBAS™ Taqman™ automated HCV test (v2.0 assay) used in this study has a LLoQ of 15 IU/mL.
Time Frame: TW4, TW8, and TW12
Population: The subset of the FAS population consisting of all participants treated with any study medication in Arms 1, 2, and 3 and who had undetectable HCV RNA at Week 4, Week 8, or Week 12.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm 1: 16-week Treatment Arm | Arm 2: 28-week Treatment Arm | Arm 3: 48-week Treatment Arm
Number analyzed (Participants) | 102 | 105 | 20
Percentage of Participants
  % Undetectable HCV RNA at TW4 (n=25, 18, 0) | 24.5 | 14.3 | 0.0
  % Undetectable HCV RNA at TW8 (n=101, 104, 0) | 69.6 | 81.0 | 0.0
  % Undetectable HCV RNA at TW12 (n=100, 103, 20) | 68.6 | 80.0 | 41.4

4. Secondary Outcome: Percentage of Participants With Relapse
Description: The percentage of viral relapse (defined as confirmed HCV RNA >15 IU/mL after End-of-Treatment [EOT]) among participants who had undetectable HCV RNA at EOT was determined for each arm. The Roche COBAS™ Taqman™ automated HCV test (v2.0 assay) used in this study has a LLoQ of 15 IU/mL.
Time Frame: From EOT to FW12 (up to 12 weeks)
Population: Participants in the FAS with undetectable HCV RNA at EOT and who have data available at FW12 were included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm 1: 16-week Treatment Arm | Arm 2: 28-week Treatment Arm | Arm 3: 48-week Treatment Arm
Number analyzed (Participants) | 93 | 90 | 18
Percentage of Participants | 20.4 | 1.1 | 0.0

5. Secondary Outcome: Percentage of Participants With Neutropenia
Description: The percentage of participants with neutropenia (neutrophil count <0.75 x10^9/L) is summarized for each arm.
Time Frame: Up to 60 weeks
Population: The All Participants as Treated (APaT) includes all participants who received ≥1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Groups:
- Arm 3: 48-week Treatment Arm: After completing the 12-week lead-in, participants with detectable HCV RNA were allocated to receive an additional 24 weeks of BOC + PR and an additional 12 weeks of PR, for a total of 48 weeks of treatment. At Week 48, participants underwent 12 weeks of follow-up (participation complete at Week 60). In addition, 21 participants who were treated but discontinued prior to Week 12 are included in Arm 3 for safety analyses.
Arm/Group | Arm 1: 16-week Treatment Arm | Arm 2: 28-week Treatment Arm | Arm 3: 48-week Treatment Arm
Number analyzed (Participants) | 102 | 105 | 50
Percentage of Participants | 10.8 | 12.4 | 4.0

6. Secondary Outcome: Percentage of Participants With Anemia
Description: The percentage of participants with anemia (hemoglobin [Hgb] <10 g/dL) was determined in each arm.
Time Frame: Up to 60 weeks
Population: The All Participants as Treated (APaT) includes all participants who received ≥1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm 1: 16-week Treatment Arm | Arm 2: 28-week Treatment Arm | Arm 3: 48-week Treatment Arm
Number analyzed (Participants) | 102 | 105 | 50
Percentage of Participants | 33.3 | 43.8 | 26.0

7. Secondary Outcome: Percentage of Participants With Dose Discontinuation Due to Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. The percentage of participants who discontinued from BOC, BOC + RBV, or all medications due to an AE are reported.
Time Frame: From TW1 through TW48
Population: The APaT includes all participants who received ≥1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm 1: 16-week Treatment Arm | Arm 2: 28-week Treatment Arm | Arm 3: 48-week Treatment Arm
Number analyzed (Participants) | 102 | 105 | 50
Percentage of Participants
  Discontinued from BOC | 2.9 | 7.6 | 16.0
  Discontinued from BOC + R | 0.0 | 5.7 | 8.0
  Discontinued from all Study Medication | 0.0 | 5.7 | 8.0

8. Secondary Outcome: Percentage of Participants With Treatment-Related Serious AEs (SAEs)
Description: A SAE is any AE that results in death, is life threatening, results in persistent or significant disability, results in or prolongs an existing inpatient hospitalization, is a congenital birth defect, is a cancer, is associated with an overdose, or is another important medical event.
Time Frame: Up to 60 weeks
Population: The APaT includes all participants who received ≥1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm 1: 16-week Treatment Arm | Arm 2: 28-week Treatment Arm | Arm 3: 48-week Treatment Arm
Number analyzed (Participants) | 102 | 105 | 50
Percentage of Participants | 2.9 | 3.8 | 4.0

ADVERSE EVENTS:
Time Frame: Up to 60 weeks
Description: A AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Arm/Group | Arm 1: 16-week Treatment Arm | Arm 2: 28-week Treatment Arm | Arm 3: 48-week Treatment Arm
Serious Adverse Events (participants affected / at risk) | 9/102 | 6/105 | 4/50
Other Adverse Events (participants affected / at risk) | 96/102 | 98/105 | 46/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: 16-week Treatment Arm (N=102) | Arm 2: 28-week Treatment Arm (N=105) | Arm 3: 48-week Treatment Arm (N=50)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucinations, mixed (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: 16-week Treatment Arm (N=102) | Arm 2: 28-week Treatment Arm (N=105) | Arm 3: 48-week Treatment Arm (N=50)
Anaemia (Blood and lymphatic system disorders) | 33 (35) | 44 (46) | 12 (13)
Neutropenia (Blood and lymphatic system disorders) | 11 (15) | 13 (15) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 8 (10) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 13 (13) | 6 (6)
Mouth ulceration (Gastrointestinal disorders) | 6 (6) | 6 (8) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (16) | 15 (15) | 11 (13)
Vomiting (Gastrointestinal disorders) | 10 (10) | 10 (11) | 6 (10)
Asthenia (General disorders) | 7 (7) | 7 (7) | 7 (7)
Chills (General disorders) | 5 (5) | 5 (5) | 8 (9)
Fatigue (General disorders) | 13 (15) | 16 (34) | 6 (20)
Influenza like illness (General disorders) | 5 (5) | 10 (26) | 5 (9)
Injection site pruritus (General disorders) | 4 (4) | 11 (12) | 0 (0)
Injection site rash (General disorders) | 5 (5) | 6 (6) | 3 (3)
Pain (General disorders) | 6 (7) | 4 (4) | 5 (5)
Pyrexia (General disorders) | 23 (48) | 23 (74) | 17 (48)
Haemoglobin decreased (Investigations) | 4 (4) | 7 (7) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 5 (5) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 18 (18) | 24 (25) | 12 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (11) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 23 (27) | 22 (31) | 7 (10)
Dizziness (Nervous system disorders) | 17 (18) | 25 (29) | 9 (12)
Dysgeusia (Nervous system disorders) | 15 (15) | 23 (24) | 8 (9)
Headache (Nervous system disorders) | 17 (18) | 18 (22) | 8 (21)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 3 (3) | 12 (12) | 0 (0)
Insomnia (Psychiatric disorders) | 16 (16) | 17 (19) | 4 (4)
Irritability (Psychiatric disorders) | 3 (3) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 14 (15) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 23 (23) | 34 (35) | 8 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 10 (11) | 6 (7)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 9 (9) | 2 (2) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 18 (19) | 4 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 6 (7) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.